CLINICAL TRIAL: NCT07250854
Title: The Use of Near-Infrared Fluorescence Cholangiography With Indocyanine Green (ICG) in the Work Up of Neonatal Cholestasis
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Sam Hagman, Fellow, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-30015542; UAB (Other: UAB)
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-11

CONDITIONS: Biliary Atresia; Kasai; Cholestasis in Newborn; Cholestasis in Newborn Infant
Keywords: biliary atresia; kasai; cholestasis; cholestasis in neonate; cholestasis in newborn; direct bilirubin; acholic stool
MeSH Terms: conditions — Biliary Atresia; Cholestasis | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cholestatic infants (Experimental): infants that are cholestatic needing further work up for biliary atresia
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — Optical imaging agent
  Other Names: ICG

SUMMARY:
In infants that present with findings concerning for biliary atresia, along with other cholestatic work up which is standard, they will receive a one-time intravenous (IV) dose of Indocyanine Green (ICG). The infant's diapers will subsequently be examined for presence of the ICG, and if present, suggests bile flow. This was described as 97% accurate for assessing biliary patency and we would like to perform a similar study to assess biliary patency in the work up of neonatal cholestasis.

ELIGIBILITY:
Inclusion Criteria:

* Infants admitted to the hospital (no matter their age, sex, race/ethnicity) who a hepatologist deems warrants inpatient work up of neonatal cholestasis suspected to be due to biliary atresia.

Exclusion Criteria:

* Infants that a hepatologist has not deemed to warrant inpatient admission for work up of neonatal cholestasis suspected to be due to biliary atresia.
* Infants that are managed in the outpatient setting
* Non-cholestatic infants
* Patient who are on TPN AND NPO for reasons other than temporary imaging or surgical requirements
* Infant with a history of bowel resection or other surgical procedures known to introduce blood into the gastrointestinal tract.

Ages: 2 Weeks to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
The number and accuracy of ICG fluorescence in the diagnosis of biliary atresia | Within 72 hours
  Measuring stool fluorescence using near infrared imaging

CONTACTS AND LOCATIONS:
Overall Officials: Laura Stafman, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama At Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No